CLINICAL TRIAL: NCT03774173
Title: A Randomised, Open-label Study to Compare Plasma Concentrations of Aramchol in Healthy Volunteers After Once or Twice Daily Oral Dosing to Steady State
Brief Title: Comparison of Aramchol Concentrations With Once or Twice Daily Dosing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galmed Pharmaceuticals Ltd (Industry)
Collaborators: Hammersmith Medicines Research (Other); Analyst Research Laboratories (Other); Diamond Pharma Services Regulatory Affairs Consultancy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Aramchol 017
Record Dates: First submitted 2018-11-29; First posted 2018-12-12 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Healthy
MeSH Terms: interventions — aramchol

STUDY DESIGN:
Intervention Model Description: Subjects will receive oral doses of aramchol at 300 mg twice daily (every 12 h) for 9 days in one period, with a single dose in the morning of Day 10, and 600 mg once daily (every 24 h) for 10 days in the other period.
  Enrolment of 16 subjects is planned with each subject taking part in the 2 study periods. The subjects will be randomised 1:1 so that 8 subjects receive each regimen in the first period and the alternate regimen in the second period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Aramchol 300 mg (Experimental): Aramchol 300 mg twice daily (every 12 hours)
  Interventions: Drug: Aramchol
- Aramchol 600 mg (Experimental): Aramchol 600 mg once daily (every 24 hours)
  Interventions: Drug: Aramchol

INTERVENTIONS:
Drug: Aramchol — One Aramchol tablet (300 mg) twice daily and 2 Aramchol tablets (300 mg each) once daily

SUMMARY:
The trial is an open-label, 2-period, randomised, crossover study of the plasma concentrations of aramchol, in which subjects will receive oral doses of aramchol at 300 mg twice daily and 600 mg once daily.

DETAILED DESCRIPTION:
The trial is an open-label, 2-period, randomised, crossover study of the plasma concentrations of aramchol, in which subjects will receive oral doses of aramchol at 300 mg twice daily (every 12 h) for 9 days in one period, with a single dose in the morning of Day 10, and 600 mg once daily (every 24 h) for 10 days in the other period. A pharmacokinetic profile will be obtained over the dosing interval on Day 10 of each period.

Enrolment of 16 subjects is planned with each subject taking part in the 2 study periods. The subjects will be randomised 1:1 so that 8 subjects receive each regimen in the first period and the alternate regimen in the second period.

Subjects will be screened within 21 days before their first dose of study medicine. In each period they will remain resident on the ward from Day -1 until the morning of Day 11. Subjects will attend a follow-up visit 14 days (±2 days) after the end of the second period. There will be an interval of at least 7 days between Periods 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female healthy volunteer.
2. Aged 18-45 years at time of consent.
3. A body mass index (BMI; Quetelet index) in the range 18.0-30.9.
4. Ability to understand the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of, the entire trial.
5. Willingness to give written consent to participate after reading and understanding the information and consent form, and after having the opportunity to discuss the trial with the investigator or his delegate.
6. Agree to use effective contraception as described in Section 11.
7. Agree not to donate blood or blood products during the study and for up to 3 months after the administration of the trial medication.
8. Willingness to give written consent to have data entered into The Overvolunteering Prevention System (TOPS).

Exclusion Criteria:

1. Woman who is pregnant or lactating, or pre-menopausal woman who is sexually active and not using a reliable method of contraception (see Section 11).
2. Of East Asian descent including, but not limited to, Chinese, Japanese, Korean, Mongolian, or Vietnamese.
3. Smoker, or has smoked cigarettes or other tobacco or nicotine products in the last 12 months.
4. Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the pre-trial screening assessment that could interfere with the objectives of the trial or the safety of the volunteer.
5. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) or alkaline phosphatase (AP) >ULN at the screening visit. A repeat is allowed on one occasion for determination of eligibility.
6. Presence of acute or chronic illness or history of chronic illness sufficient to invalidate the volunteer's participation in the trial or make it unnecessarily hazardous.
7. History or presence of any disease or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs including gastrointestinal disorder or of oesophageal, gastric, biliary or intestinal surgery (excluding herniotomy and appendectomy).
8. Use of anticholinergic or other drugs known to affect gastrointestinal motility during the 7 days before the first dose of trial medication.
9. Impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease, or history of any psychotic mental illness.
10. Surgery (eg stomach bypass) or medical condition that might affect absorption of medicines.
11. Presence or history of severe adverse reaction to any drug or a history of sensitivity to aramchol, cholic acid, bile acid sequestrants, or any excipients in the tablets.
12. Use of a prescription medicine (except oral contraceptives in females), or any other medicine or herbal remedy (including St John's wort) known to interfere with enzymes in the liver, during the 28 days before the first dose of trial medication; or use of any other over-the-counter medicine, with the exception of acetaminophen (paracetamol), during the 7 days before the first dose of trial medication.
13. Receipt of an investigational product (including prescription medicines) as part of another clinical trial within the 3 months before first admission to this study; in the follow-up period of another clinical trial at the time of screening for this study.
14. Presence or history of drug or alcohol abuse, or intake of more than 14 units of alcohol weekly.
15. Blood pressure and heart rate in supine position at the screening examination outside the ranges: blood pressure 100-140 mm Hg systolic, 50-90 mm Hg diastolic; heart rate 45_90 beats/min, unless judged not clinically significant. Borderline values (ie values that are within 5 mm Hg for blood pressure or 5 beats/min for heart rate) will be repeated. Subjects can be included if the repeat value is within range or still borderline, but deemed not clinically significant by the investigator.
16. Possibility that the volunteer will not cooperate with the requirements of the protocol.
17. Evidence of drug abuse on urine testing.
18. Positive test for hepatitis B, hepatitis C or HIV.
19. Loss of more than 400 mL blood during the 3 months before the trial, eg as a blood donor.
20. Objection by GP to volunteer entering trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-12-08 (Actual); Primary Completion 2019-02-03 (Actual); Study Completion 2019-03-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of aramchol | PK parameters will be measured on Days 7, 8 , 9, and 10.
  AUC
Pharmacokinetics of aramchol | PK parameters will be measured on Days 7, 8 , 9, and 10.
  Cavg
PK of aramchol | PK parameters will be measured on Days 7, 8 , 9, and 10.
  Ctau
Pharmacokinetics (PK) of aramchol | K parameters will be measured on Days 7, 8 , 9, and 10.
  Tmax

SECONDARY OUTCOMES:
Vital signs and physical examination | During both treatment periods vital signs will be assessed on Days 1, 5 and 10.
  Systolic and diastolic blood pressure, Heart rate, Oral temperature and Respiratory rate
Electrocardiogram | During both treatment periods ECG will be assessed on Days 1, 5 and 10.
  12-lead ECGs
Laboratory safety tests: Biochemistry | On Day -1, Day 5,on Day 11.
  Usual tests.
Laboratory safety tests: Hematology | On Day -1, Day 5,on Day 11.
  haemoglobin, red blood cells, mean corpuscular volume , mean corpuscular haemoglobin, mean corpuscular haemoglobin concentration, haematocrit, white blood cells and platelets.
Laboratory safety tests: Urinalysis | On Day -1, Day 5,on Day 11.
  Usual Dipstick test
Safety and tolerability: Adverse events (AEs). | From screening visit to 14 days after the last dose in period 2.
  Adverse events are collected during entire study period.

CONTACTS AND LOCATIONS:
Overall Officials: Adeep Puri, M.D., Principal Investigator — Hammersmith Medicines Research
Locations (1):
- Hammersmith Medicines Research (HMR), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No